CLINICAL TRIAL: NCT05715203
Title: Aortic Stiffness in Patients With Genetic Aortopathies: Intervention Analysis
Brief Title: Aortic Stiffness in Patients With Genetic Aortopathies
Acronym: PULSEWAVE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: Pulse Wave
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Rare Diseases; Aortic Stiffness; Connective Tissue Defect
Keywords: arterial stiffness; Ascending aortic aneurysm; pulse wave velocity
MeSH Terms: conditions — Rare Diseases; Aneurysm, Ascending Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Syndromic TAA: Subjets with clinical or genetic diagnosis of syndromic thoracic aortic aneurysms
  Interventions: Device: Pulsotonometry
- Non-syndromic TAA: Subjets without clinical or genetic diagnosis of syndromic thoracic aortic aneurysms
  Interventions: Device: Pulsotonometry

INTERVENTIONS:
Device: Pulsotonometry — Evaluation of arterial stiffness

SUMMARY:
The goal of this observational study is to study arterial stiffness in patients with thoracic ascending aortic aneurysms (TAA), either syndromic or non-syndromic. The main questions it aims to answer are:

* Stratification of aortic risk based on arterial stiffness; Compare measurements with morphological and haemodynamic features of the ascending thoracic aorta.

Participants will be asked to undergo non-invasive evaluation of blood pressure and arterial stiffness.

DETAILED DESCRIPTION:
Recent studies have highlighted the role played by the aorta and the great arteries in the regulation of the blood pressure (BP) and peripheral blood flow. Similarly, the structural and functional alteration of the aortic wall having a genetic cause is highly associated with the onset of aneurysms, especially of the ascending aorta, for which it is essential to monitor the aortic stiffness, which is detectable through a non-invasive and non-radioactive method such as Pulse Wave Velocity (PWV). Despite literature studies correlating PWV in MFS, few evaluations of aortic stiffness in patients with syndromic TAA have been done and its potential correlations with other aneurysm markers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with AAT, either syndromic or non syndromic;
* Signed informed consent

Exclusion Criteria:

* Patients with early menopause and/or osteoporosis, rheumatic heart disease and active malignant tumours;
* Patients with acute and chronic inflammatory conditions such as: chronic liver disease, chronic renal insufficiency and diseases affecting the thyroid system;
* Seropositivity to HIV, HCV, HBsAg and SARS-CoV-2;
* Pregnancy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ascending aortic aneurysms currently in follow.up at Cardiovascular Gentic Centre, IRCCS Policlinico San Donato.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity | 18 months
  Statistic analysis will be performed using the Statistical Package for Social Science (SPSS for Windows; v20.0; SPSS, Chicago, Illinois, USA). Continuous variables will be expressed as mean ± Standard Deviation, while qualitative variables will be expressed as a percentage. Qualitative data will be compared using Fisher's test or Pearson's χ2 test, when appropriate. Continuous variables by t-test or analysis of variance normalized for covariates. Continuous variables will be correlated by simple or multiple linear regression

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pini, Principal Investigator — Cardiovascular-Gentic Centre, IRCCS Policlinico San Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy